CLINICAL TRIAL: NCT04789356
Title: Phase IV Study to Evaluate the Effectiveness of the Inactivated Adsorbed Vaccine Against COVID-19 CoronaVac, Among Public Safety and Education Workers With Risk Factors for Severity, in Manaus (Amazonas)
Brief Title: Effectiveness of the Adsorbed Vaccine COVID-19 (Coronavac) Among Education and Public Safety Workers With Risk Factors for Severity
Acronym: COVACMANAUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 44076721.5.0000.0005
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Brazil; Covid-19; Vaccine; Sinovac; CoronaVac; Vaccine efficacy
MeSH Terms: conditions — COVID-19 | interventions — Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-risk individuals (with comorbidities) (Active Comparator): Public safety and security (police officers and law enforcement, fire department), and high school and college/university professionals of the state government public education network who present at least one of the comorbidities included in the National Plan for the Operationalization of Vaccination Against COVID-19 will be invited to receive the CoronaVac vaccine
  Interventions: Biological: Adsorbed SARS-CoV-2 (inactivated) vaccine
- Low-risk individuals (without comorbidities) (No Intervention): Participants with low risk (without comorbidities as a risk factor for severe COVID-19 according to the national plan for the implementation of vaccination against COVID-19) will not receive the vaccine within the scope of the research project.

INTERVENTIONS:
Biological: Adsorbed SARS-CoV-2 (inactivated) vaccine — 600 SU/dose; Two doses separated by 28 days (± 7 days). Intramuscular (deltoid) administration.
  Other Names: CoronaVac
  Arms: High-risk individuals (with comorbidities)

SUMMARY:
This is a quasi-experimental study with risk-based allocation. Public security and education professionals from the state government will be included. In the initial evaluation, the presence of comorbidities associated with an increased risk of serious disease due to COVID-19 will be evaluated, according to the national plan for the implementation of vaccination against COVID-19. Those with at least one of these comorbidities will be invited to receive the study vaccine in two doses, with an interval of 28 days (±7 days). Participants with low risk (without comorbidities as a risk factor for severe COVID-19 according to the national plan for the implementation of vaccination against COVID-19) will not receive the vaccine within the scope of the research project. If, after 12 months, the participant in the low-risk group (no vaccine) has not received CoronaVac, or any other vaccine available, he/she will receive the vaccine, exactly as offered in the other group (two doses of CoronaVac with an interval of 28 days - with a tolerance of 7 days before or after). All participants will be followed up for 12 months from inclusion in the study. Immunization is expected to reduce the risk of moderate to severe disease of those with comorbidities to the level of those of the same age group who do not have these comorbidities but face similar occupational risks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 49 years
* Demonstrate availability to be accompanied during the follow-up time defined in the study, through visits, telephone contacts, or other means of digital communication.

Exclusion Criteria:

* Prior vaccination for COVID-19;
* Diagnosis of COVID-19 in the last 28 days (nasal and oropharyngeal swab);
* History of severe allergic reaction or anaphylaxis to study vaccine components;
* Report of fever in the 72 hours prior to vaccination (the inclusion may be postponed until the participant completes 72 hours without fever);
* Possible or confirmed of COVID-19 on the day of vaccination (in this situation, vaccination can be postponed until the participant completes 72 hours without symptoms or the diagnosis is ruled out);
* Have received live attenuated virus vaccine in the last 28 days or inactivated vaccine in the last 14 days prior to inclusion in the study, or have immunization scheduled for the first 28 days after their inclusion in the study;
* Any other condition that, in the opinion of the principal investigator or his medical representative, could endanger the safety or rights of a potential participant or that would prevent him or her from complying with this protocol;
* Pregnancy or breastfeeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6233 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Incidence density of moderate and severe clinical cases of COVID-19 | 2 weeks after the second vaccine dose
  Incidence density of moderate and severe clinical cases of COVID-19 (Grade 4 or higher according to the WHO clinical progression scale), after the second week after the second dose of the vaccine.

SECONDARY OUTCOMES:
Incidence density of moderate and severe clinical cases of COVID-19 after first dose | After first dose, up to 12 months.
  Incidence density of moderate and severe clinical cases of COVID-19 (grade 4 or higher according to the WHO clinical progression scale) from the first dose
Incidence density of moderate and severe clinical cases of COVID-19 after second dose | After second dose, up to 12 months.
  Incidence density of moderate and severe clinical cases of COVID-19 (grade 4 or higher according to the WHO clinical progression scale) from the second dose
Incidence density of severe clinical cases of COVID-19 after second dose | After second dose, up to 12 months.
  Incidence density of severe clinical cases of COVID-19 (grade 6 or higher according to the WHO clinical progression scale) from the second dose
Median of clinical progression scores between moderate and severe cases | After first dose, up to 12 months.
  Comparison of the median clinical progression scores according to the WHO clinical progression scale between groups
Incidence density of clinical cases virologically confirmed as COVID-19 | After first dose, up to 12 months.
Mortality confirmed as COVID-19 | After first dose, up to 12 months.
  Incidence density of deaths confirmed as COVID-19
Incidence density of hospitalizations for any cause | After first dose, up to 12 months.
Mortality from any cause | After first dose, up to 12 months.
  Density of mortality from any cause
Adverse events | Up to 7 days after each dose of the vaccine (Day 7 and Day 35)
  Frequency of adverse events associated with the need for medical care
Humoral and cell-mediated immune response | Before each vaccine dose and every 3 months, up to 12 months of follow-up.
  Quantification of humoral and cell-mediated immune response to vaccination in samples of a subgroup of participants
Detection of antibodies against SARS-CoV-2 in samples | Before each vaccine dose and every 3 months, up to 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lacerda, MD, Principal Investigator — Fundação de Medicina Tropical Heitor Vieira Dourado
Locations (1):
- Escola Normal Superior - Universidade do Estado do Amazonas, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided